CLINICAL TRIAL: NCT04617717
Title: Personalized Treatment for Patients With Premature Ventricular Beats
Status: Recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Mathis Korseberg Stokke, Professor and Consultant Cardiologist, Oslo University Hospital
Other Study IDs: 153850
Record Dates: First submitted 2020-10-26; First posted 2020-11-05 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Ventricular Premature Complexes
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Exercise Test; Electrocardiography, Ambulatory; Echocardiography; Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Invasive cardiac electrophysiological study and ablation therapy — Invasive cardiac electrophysiological study with cathecholamine provocation and pacing procedures, as well as standard 3D mapping and PVC ablation
Diagnostic Test: Cardiopulmonary exercise testing — Standard ergometer bicycle test
Diagnostic Test: Cardiac MRI — Cardiac MRI with cine-imaging and late-gadolinium enhancement
Diagnostic Test: Holter monitoring — 24h 5 lead or 12 lead ECG recording
Diagnostic Test: Transthoracic echocardiography — 2D echocardiography
Diagnostic Test: Coronary angiography — Conventional invasive coronary angiography or CT angiography as indicated

SUMMARY:
Frequent premature ventricular beats (PVBs) are common, negatively affects the quality of life for many patients, and can lead to impaired contractile function. Rule-out of structural heart disease is key in the assessment of PVBs. Cardiac MR has a high sensitivity for structural heart disease, but the diagnostic gain from this resource-demanding procedure in the work-up of patients with PVBs is unknown. There is a need to establish the role of MR in the evaluation of patients with PVBs to improve diagnostic efficacy, establish treatment strategies, and promote further research. This project will answer three key questions: 1) What is the diagnostic gain from cardiac MR in patients with PVBs? 2) Is MR the real gold standard to rule-out structural heart disease in patients with PVBs? 3) Can non-invasive heart rate parameters guide the strategy for induction of PVBs during invasive electrophysiological procedures?

ELIGIBILITY:
Inclusion Criteria: Patients referred for PVC ablation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to PVC ablation
Sampling Method: Non-Probability Sample
Enrollment: 224 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2040-07-31 (Estimated)

PRIMARY OUTCOMES:
MRI-based evidence of structural heart disease | 3-5 years
  Evidence of structural heart disease from MRI compared to echocardiography
PVC induction vs PVC/HR-relationship | 3-5 years
  Correlation of method for induction of PVCs during invasive procedure vs PVC/HR relationship during CPET
EPS-based evidence of structural heart disease | 3-5 years
  Evidence of structural heart disease from invasive electrophysiology vs MRI and echo

CONTACTS AND LOCATIONS:
Overall Officials: Mathis K Stokke, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No